CLINICAL TRIAL: NCT03151876
Title: Chidamide Combined With Cladribine/Gemcitabine/Busulfan (ChiCGB) With Autologous Stem-Cell Transplantation in Relapsed and Refractory Diffuse Large B Cell Lymphoma
Brief Title: Chidamide Combined With Clad/Gem/Bu With AutoSCT in R/R Diffuse Large B Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Clinical Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChiCGB-DLBCL
Record Dates: First submitted 2017-05-05; First posted 2017-05-12 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Cladribine; Gemcitabine; Busulfan

STUDY DESIGN:
Intervention Model Description: ChiCGB
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ChiCGB (Experimental): Experimental: ChiCGB
  Chidamide administered orally on D-7, -4, 0,+3
  Cladribine administered at 10mg on D-6 to D-2
  Gemcitabine administered at 2500 mg/m2 on days -6 and -2.
  Busulfan administered at 3.2 mg/kg (adjusted ideal body weight) on days -6 to -3.
  Dexamethasone 10 mg by vein daily from day -6 to day -1. Caphosol oral rinses 30 mL four times a day used from day -8.
  Interventions:
  Drug: Chidamide Drug: Cladribine Drug: Gemcitabine Drug: Busulfan Drug: Dexamethasone Procedure: Stem Cell Transplant
  Interventions: Drug: Chidamide; Drug: Cladribine; Drug: gemcitabine; Drug: Busulfan; Procedure: Autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: Chidamide — 30 mg oral twice weekly for 2 weeks
Drug: Cladribine — 6 mg/m2 intravenously daily for 5 days
Drug: gemcitabine — 2500 mg/m2 intravenously twice weekly for 1 week
Drug: Busulfan — 3.2 mg/kg intravenously daily for 4 days
Procedure: Autologous hematopoietic stem cell transplantation — autologous hematopoietic stem cells infusion after ChiCGB chemotherapy

SUMMARY:
The goal of this clinical research study is to evaluate effectiveness and safety of ChiCGB regimen( chidamide, cladribine, gemcitabine and busulfan).

Busulfan are designed to kill cancer cells by binding to DNA (the genetic material of cells), which may cause cancer cells to die.

Gemcitabine and cladribine are designed to disrupt the growth of cancer cells, which may cause cancer cells to die. It may help to increase the effect of busulfan on cancer cells by not allowing these cells to repair the DNA damage caused by busulfan.

Chidamide is designed to open up the DNA and allow greater access to drugs that bind to DNA, such as cladribine, gemcitabine, busulfan.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be enrolled in a group of at least 3 participants to begin receiving the study drugs.

The dose of the study drugs you receive will depend on when you enrolled in this study. If no intolerable side effects occur in your group, researchers will continue to enroll participants at the next dose level until either the vorinostat reaches the dose level currently used alone without stem cell transplant, or the highest tolerable dose of this drug is found. The dose that you receive will remain the same throughout this study.

You will be admitted to the hospital on Day -6.

Study Drug Administration (for all patients):

In stem cell transplant, the days before you receive your stem cells are called minus days. The day you receive the stem cells is called Day 0. The days after you receive your stem cells are called plus days.

On Day -7, -4, 0, +3 , you will take chidamide by mouth.

On Days -6, -5, -4, -3, and -2 you will receive cladribine by vein over 1/2 hours.

On Day -6, -2, you will receive gemcitabine by vein over 3 1/2 - 4 1/2 hours.

On Days -6, -5, -4, and -3, you will receive busulfan by vein over 3 hours.

On Day -1, you will rest.

On Day 0, you will receive your stem cells by vein over about 30-60 minutes.

As part of standard care, you will receive G-CSF (filgrastim) as an injection just under your skin twice a day starting on Day +5 until your blood cell levels return to normal.

Study Tests:

On Day -1, you will have an electrocardiogram (ECG) to check your heart function.

About 30-100 days after the transplant, you will have lung function tests.

About 100 days after the transplant:

Blood (about 4 teaspoons) will be drawn for routine tests. If the doctor thinks it is needed, you may have a bone marrow aspiration and biopsy to check the status of the disease.

You will have a PET/CT scan of your whole body to check the status of the disease.

Length of Study:

As part of standard care, you will remain in the hospital for about 3-4 weeks after the transplant. After you are released from the hospital, you will continue as an outpatient for infections and transplant-related complications.

You will be taken off study about 100 days after the transplant. You may be taken off study early if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

This is an investigational study. Chidamide, gemcitabine, busulfan, melphalan, and rituximab are all FDA approved and commercially available. The use of these study drugs in combination is investigational.

Up to 93 patients will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary refractory or recurrent diffuse large B cell lymphoma that do not qualify for treatment protocols of higher priority.
2. Relapsed patients should respond to 2nd or 3rd line salvage chemotherapy and attain at least PR before recruitment.
3. Adequate renal function, as defined by estimated serum creatinine clearance >/=50 ml/min and/or serum creatinine </= 1.8 mg/dL.

6. Adequate hepatic function, as defined by serum glutamate oxaloacetate transaminase (SGOT) and/or serum glutamate pyruvate transaminase (SGPT) </= 3 x upper limit of normal; serum bilirubin and alkaline phosphatase </= 2 x upper limit of normal.

7. Adequate pulmonary function with forced expiratory volume at one second (FEV1), forced vital capacity (FVC) and diffusing capacity of lung for carbon monoxide (DLCO) >/= 50% of expected corrected for hemoglobin.

8. Adequate cardiac function with left ventricular ejection fraction >/= 50%. No uncontrolled arrhythmias or symptomatic cardiac disease.

9. Performance status 0-1. 10. Negative Beta diffusing capacity of lung for carbon monoxide (HCG) text in a woman with child-bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization

Exclusion Criteria:

1. Central nervous system lymphoma
2. Patients relapsed after ASCT
3. Bone marrow was involved by lymphoma
4. Patients with active hepatitis B or C(HBV DNA >/=10,000 copies/mL).
5. Active infection requiring parenteral antibiotics
6. HIV infection, unless the patient is receiving effective antiretroviral therapy with undetectable viral load and normal cluster of differentiation 4 (CD4) counts
7. Evidence of either cirrhosis or stage 3-4 liver fibrosis in patients with chronic hepatitis C or positive hepatitis C serology.
8. Patients with a cQT longer than 500 ms

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 2 years

SECONDARY OUTCOMES:
Overall survival | 2 years
Complete remission | 3 month after autologous hematopoietic stem cell transplantation
Adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ting Liu, MD, Principal Investigator — West China Hospital
Locations (18):
- China (18):
  - Beijing cancer hospital, Beijing, Beijing Municipality
  - Peking university third hospital, Beijing, Beijing Municipality
  - The first affiliated hospital of Chongqing medical university, Chongqing, Chongqing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - General Hospital of Lanzhou military command, Lanzhou, Gansu
  - Henan cancer hospital, Zhengzhou, Henan
  - The first affiliated hospital of Zhengzhou university, Zhengzhou, Henan
  - Tongji Hospital, Wuhan, Hubei
  - Jiangsu province hospital, Nanjing, Jiangsu
  - Rui jin hospital Shanghai jiao tong University, Shanghai, Shanghai Municipality
  - Tong Ren Hospital, Shanghai, Shanghai Municipality
  - Shan Xi Da Yi Hospital, Taiyuan, Shanxi
  - Tangdu Hospital, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital of Southwest Medical University, Nanchong, Sichuan
  - Blood diseases hospital, Chinese academy of medica, Tianjin, Tianjing
  - The first affiliated hospital of Xinjiang medical Universtiy, Ürümqi, Xinjiang
  - Kunming General Hospital of Chengdu Military Area, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Yes
electronic case report form (eCRF)

REFERENCES:
- [Derived] Ji J, Liu Z, Kuang P, Dong T, Chen X, Li J, Zhang C, Liu J, Zhang L, Shen K, Liu T. A new conditioning regimen with chidamide, cladribine, gemcitabine and busulfan significantly improve the outcome of high-risk or relapsed/refractory non-Hodgkin's lymphomas. Int J Cancer. 2021 Dec 15;149(12):2075-2082. doi: 10.1002/ijc.33761. Epub 2021 Aug 25. PMID 34398971